CLINICAL TRIAL: NCT01085929
Title: Ultrasound Guided Needle Drainage Versus Formal Incision and Drainage of Superficial Soft Tissue Abscesses in the Emergency Department Setting
Brief Title: Incision and Drainage Versus Needle Aspiration in Soft Tissue Abscesses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Romolo Gaspari, University of Massachusetts
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UMass12522
Record Dates: First submitted 2010-03-10; First posted 2010-03-12 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2010-03

CONDITIONS: Abscess; Cellulitis
Keywords: abscess; infection; ultrasound guidance; incision and drainage; needle aspiration; skin; ultrasound
MeSH Terms: conditions — Abscess; Cellulitis; Infections; Surgical Wound | interventions — Drainage; Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Incision and Drainage (Active Comparator): Abscess underwent incision and drainage
  Interventions: Procedure: Incision and Drainage
- Ultrasound guided needle aspiration (Active Comparator): Ultrasound was used to identify the abscess location. A needle was introduced into the abscess cavity and aspiration of the contents were attempted.
  Interventions: Procedure: Ultrasound Guided Aspiration

INTERVENTIONS:
Procedure: Incision and Drainage — Surgical incision of the skin surface followed by expression of purulence with or without debridement or manual exploration of abscess cavity.
  Arms: Incision and Drainage
Procedure: Ultrasound Guided Aspiration — Ultrasound is used to identify the abscess cavity. An 18 gauge needle is introduced into the abscess cavity and manual aspiration of the abscess contents is attempted.
  Arms: Ultrasound guided needle aspiration

SUMMARY:
The incidence of skin and soft tissue infections has increased dramatically over the last decade, in part due to increased prevalence of community-acquired methicillin-resistant Staphylococcus aureus (CA-MRSA). Incision and drainage (I&D) is considered the primary intervention, however some clinicians prefer ultrasound guided needle aspiration (US Asp). The investigators performed a randomized trial comparing US Asp to I&D for uncomplicated skin and soft tissue abscesses, with a subgroup analysis of patients with CA-MRSA.

ELIGIBILITY:
Inclusion Criteria:

* presenting to emergency department with skin abscess
* abscess required surgical drainage
* healthy appearing

Exclusion Criteria:

* pregnant
* unable to give consent
* abscess located in oral cavity
* abscess located on genitalia
* abscess located intra-gluteal at coccyx

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-08; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Successful drainage of abscess | 7 days
  Clinical outcome at 7 days

SECONDARY OUTCOMES:
Successful drainage of abscess | 2 days
  Healing of abscess following drainage procedure at day 2
Ability to evacuate purulence from abscess | Day 1
  Amount of purulence produced by drainage procedure on day 1

CONTACTS AND LOCATIONS:
Overall Officials: Romolo Gaspari, MD, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (2):
- United States (2):
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts